CLINICAL TRIAL: NCT02959112
Title: Epinephrine Sprayed on the Papilla and Rectal Indomethacin Versus Sterile Water Sprayed on the Papilla and Rectal Indomethacin for Preventing Pancreatitis After Endoscopic Retrograde Cholangiopancreatography: A Prospective, Randomized, Controlled Trial
Brief Title: Epinephrine Sprayed on the Papilla Versus Sterile Water Sprayed on the Papilla for Preventing Pancreatitis After Endoscopic Retrograde Cholangiopancreatography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because previous studies had found no difference, and one recent study even reported a higher incidence of PEP in treatment arm
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, FELIX IGNACIO TELLEZ AVILA, M.D., M.Sc., Ph. D., Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2008
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pancreatitis, Acute
Keywords: pancreatitis after ERCP; epinephrine; papilla; rectal indomethacin
MeSH Terms: conditions — Pancreatitis | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: Participants were allocated into groups by block randomisation using computed-generated numbers. The two groups were rectal indomethacin and epinephrine sprayed on the ampulla versus rectal indomethacin and sham water spray.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: As the two solutions are colourless, the endoscopist, nurse and patient were all blinded to the intervention. Investigators who participated in the evaluation of post-ERCP complications were also blinded to group allocation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epinephrine sprayed on the papilla and rectal indomethacin (Active Comparator): Epinephrine 1 mg/1 mL + 9 mL of sterile water are sprayed on the papilla at the end of the endoscopic retrograde cholangiopancreatography and 100 mg of indomethacin rectal suppository is administered at the beginning of the procedure
  Interventions: Drug: Epinephrine; Other: Sterile water; Drug: Indomethacin Rectal Suppository
- Sterile water sprayed on the papilla and rectal indomethacin (Placebo Comparator): 10 mL of sterile water are sprayed on the papilla at the end of the endoscopic retrograde cholangiopancreatography and 100 mg of indomethacin rectal suppository is administered at the beginning of the procedure
  Interventions: Other: Sterile water; Drug: Indomethacin Rectal Suppository

INTERVENTIONS:
Drug: Epinephrine
  Arms: Epinephrine sprayed on the papilla and rectal indomethacin
Other: Sterile water
Drug: Indomethacin Rectal Suppository

SUMMARY:
This multicentre randomised controlled trial included patients aged >18 years with an indication for ERCP and naive major papilla. All patients received 100 mg of rectal indomethacin and 10 ml of either sterile water or a 1:10,000 epinephrine dilution. Patients were asked about PEP symptoms via telephone 24 hours and 7 days after the procedure.

DETAILED DESCRIPTION:
This multicentre randomised placebo-controlled trial was conducted in two hospitals in Mexico: the National Institute of Medical Sciences and Nutrition "Salvador Zubirán" (INCMNSZ) in Mexico City, and Bernardette Hospital in Jalisco. The study was approved by both institutional review boards. All patients provided written informed consent.

All patients were given a dose of rectal indomethacin (100 mg) at the beginning of the ERCP. Depending on the experimental group, either 10 ml of sterile water or 10 ml of a 1:10,000 epinephrine dilution (0.1 mg/ml) was sprayed on the ampulla through a biliary balloon or a sphincterotome, avoiding any direct contact with the papilla during irrigation at the end of the procedure.

After the procedure, patients were monitored in the recovery room for 2 hours and then discharged. Symptoms of acute pancreatitis or any other complication were interrogated at baseline while in the recovery room, and then by telephone 24 hours and 7 days after the procedure. Serum levels of pancreatic enzymes were determined only if the patient developed abdominal pain after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient with an indication for endoscopic retrograde cholangiopancreatography
* Patient without prior endoscopic retrograde cholangiopancreatography
* Patient who accept contact by telephone

Exclusion Criteria:

* Previous sphincterotomy
* Allergy to epinephrine or indomethacin
* NSAIDs use in the prior week
* Pancreatic cancer located in the head
* Chronic pancreatitis
* Renal failure (Cr >1.4 mg / dl)
* Indication for endotracheal intubation independent of endoscopic retrograde cholangiopancreatography
* Biliodigestive derivation
* Pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with pancreatitis after endoscopic retrograde cholangiopancreatography, used consensus definition | 7 days
  Consensus definition for post endoscopic retrograde cholangiopancreatography pancreatitis is: (1) new or worsened abdominal pain, (2) new or prolongation of hospitalization for at least 2 days, and (3) serum amylase or lipase 3 times or more the upper limit of normal, measured more than 24 hours after the procedure

SECONDARY OUTCOMES:
Risk factors associated with the development of pancreatitis after endoscopic retrograde cholangiopancreatography assessed by relative risk | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romano-Munive AF, Garcia-Correa JJ, Garcia-Contreras LF, Ramirez-Garcia J, Uscanga L, Barbero-Becerra VJ, Moctezuma-Velazquez C, Ochoa-Rubi JA, Toledo-Cuque J, Vazquez-Anaya G, Keil-Rios D, Grajales-Figueroa G, Ramirez-Luna MA, Valdovinos-Andraca F, Zamora-Nava LE, Tellez-Avila F. Can topical epinephrine application to the papilla prevent pancreatitis after endoscopic retrograde cholangiopancreatography? Results from a double blind, multicentre, placebo controlled, randomised clinical trial. BMJ Open Gastroenterol. 2021 Feb;8(1):e000562. doi: 10.1136/bmjgast-2020-000562. PMID 33558263